CLINICAL TRIAL: NCT00165412
Title: Breast MRI Screening in Women Treated With Mediastinal Irradiation for Hodgkin's Disease
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Andrea K. Ng, MD, Radiation Oncologist, Dana-Farber Cancer Institute
Other Study IDs: 05-241
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Hodgkin's Disease
Keywords: Breast screening; Breast MRI; Mammogram; Mammography
MeSH Terms: conditions — Breast Neoplasms; Hodgkin Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: breast MRI — Repeated once a year for three years
Procedure: Mammogram — Repeated once a year for three years

SUMMARY:
The purpose of this study is to determine if the use of breast MRI in detecting breast malignancies in survivors of Hodgkin's disease is more successful than the traditional mammogram.

DETAILED DESCRIPTION:
* The screening breast MRI and mammography will be performed 6 months or longer after the last mammogram. For pre-menopausal women, the screening will be performed during the second week of the menstrual cycle to reduce cycle-related breast changes. As much as possible, the breast MRI and mammogram are to be performed on the same day.
* On the day of the breast imaging studies, the patient will also be asked to fill out a baseline breast health questionnaire, which includes questions on time since radiation therapy, prior screening history, history of prior benign breast biopsies, menopausal status, prior hormonal therapy use, etc.
* In patients with suspicious findings or findings highly suggestive of malignancy, the abnormal findings will be reviewed with the patient and recommendations will be made for a biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients treated with radiation therapy to the chest area for Hodgkin's disease
* Age between 12 and 35 at initial treatment
* Eight years or longer after initial treatment
* Pre-approval from the participant's insurance company for the breast imaging studies

Exclusion Criteria:

* Pregnant or lactating women
* Post Bilateral mastectomy
* Currently undergoing breast cancer therapy
* Known metastatic cancer
* Patients with contraindications for undergoing an MRI: cardiac pacemaker, known metallic objects in body e.g. metallic clips, bullets, shrapnel or buckshots.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Survivors of Hodgkin's disease that have been previously received radiation therapy to the chest area
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2005-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To compare the sensitivity, specificity, positive and negative predictive value of mammography and breast MRI for breast cancer detection in women treated for Hodgkin's disease. | 5 years

SECONDARY OUTCOMES:
To describe the MRI appearance and enhancing characteristics of breast cancer after Hodgkin's disease | 5 years
to correlate the breast MRI findings and pathological findings | 5 years
to determine the incidence of interval breast cancer in the screened population. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea K. Ng, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Ng AK, Garber JE, Diller LR, Birdwell RL, Feng Y, Neuberg DS, Silver B, Fisher DC, Marcus KJ, Mauch PM. Prospective study of the efficacy of breast magnetic resonance imaging and mammographic screening in survivors of Hodgkin lymphoma. J Clin Oncol. 2013 Jun 20;31(18):2282-8. doi: 10.1200/JCO.2012.46.5732. Epub 2013 Apr 22. PMID 23610104